CLINICAL TRIAL: NCT06020495
Title: Systematic Use of DDAVP to Prevent Serum Sodium Overcorrection in Severe Hyponatremia: a Multicenter Open-label Randomized Controlled Trial
Brief Title: Systematic Use of DDAVP to Prevent Serum Sodium Overcorrection in Severe Hyponatremia
Acronym: DASSOH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP220676
Record Dates: First submitted 2023-08-28; First posted 2023-08-31 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Hyponatremia
MeSH Terms: conditions — Hyponatremia | interventions — Deamino Arginine Vasopressin

STUDY DESIGN:
Intervention Model Description: Multicentre, prospective, open-label randomized controlled superiority trial with stratification on the presence of neurological symptoms at inclusion and on the presence/absence of risk factors for central pontine myelinolysis (chronic alcohol abuse, malnutrition, serum potassium < 3.0 mmol/L).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DDAVP (Experimental): DDAVP 4µg/ml IV Additional doses may be administrated every 6h for a maximum of 48h
  - Standard hyponatremia treatment : Presence of neurological symptoms : sodium chloride 3% 150ml for 20 min Absence of neurological symptoms : Hyper or isotonic fluid but never hypotonic
  Interventions: Drug: DDAVP
- Standard hyponatremia treatment (Active Comparator): Standard hyponatremia treatment alone :
  Presence of neurological symptoms : sodium chloride 3% 150ml for 20 min Absence of neurological symptoms : Hyper or isotonic fluid but never hypotonic
  Interventions: Drug: Standard hyponatremia treatment

INTERVENTIONS:
Drug: DDAVP — Posology: 4µg in 2ml IV solution Route of administration: Intravenous Duration of treatment: 48h maximum (additional doses every 6h)
  Arms: DDAVP
Drug: Standard hyponatremia treatment — Standard hyponatremia treatment alone :
  Presence of neurological symptoms :
  sodium chloride 3% 150ml for 20 min Absence of neurological symptoms : Hyper or isotonic fluid but never hypotonic
  Arms: Standard hyponatremia treatment

SUMMARY:
ICU patients with severe hyponatremia and a high risk of rapid SNa overcorrection.

DETAILED DESCRIPTION:
Multicentre, prospective, open-label randomized controlled superiority trial with stratification on the presence of neurological symptoms at inclusion and on the presence/absence of risk factors for central pontine myelinolysis (chronic alcohol abuse, malnutrition, serum potassium < 3.0 mmol/L).

Patients in ICU with severe hyponatremia defined by SNa < 115 mmol/L or SNa < 120 mmol/L in the presence of neurological symptoms (convulsions, stupor defined by a Glasgow score <12 or signs of brain herniation) and a normal or decreased extracellular fluid volume will be included.

After written informed consent, they will be randomized (1:1), using a computer-generated randomization scheme of various-sized blocks, stratified by the presence of neurological symptoms at inclusion (seizures, stupor defined as Glasgow score <12 or signs of brain herniation) and on the presence/absence of risk factors for central pontine myelinolysis (chronic alcohol abuse [defined according to World Health Organization definition], malnutrition [BMI<20.5 or weight loss >5% in 3 months], serum potassium < 3.0 mmol/L), through a centralized 24-hour Internet service (CleanWEB™), to receive standard hyponatremic treatment alone or standard hyponatremic treatment and DDAVP 4 μg/ml IV, after randomisation and for a total duration of 48 hours. Since administration of DDAVP leads to an important decrease in urine output and increase in urine osmolarity which are clinically obvious very rapidly, a single or double blind trial is not appropriate. However, all investigators will be unaware of aggregate outcomes during the study and brain MRI imaging will be performed and analyzed blinded to the randomization group

ELIGIBILITY:
Inclusion Criteria:

* Adults ( ≥18 years)
* Current admission in ICU
* Severe hyponatremia defined by SNa <120 mmol/L in the presence of neurological symptoms (seizures, stupor defined as Glasgow score < 12, or signs of brain herniation) or by SNa <115 mmol/L
* Normal or decreased extracellular fluid volume

Exclusion Criteria:

* Obvious increase of extracellular fluid volume (cirrhosis with ascites, congestive heart failure, nephrotic syndrome);
* Hyponatremia caused by hyperglycaemia (> 30 mmol/L) or hypertriglyceridemia (10 g/L) or hyperproteinaemia (120 g/L)
* Severe acute kidney injury (KDIGO 3)
* Severe chronic kidney disease (eGFR <20 ml/min)
* Coronary patients well stabilized with trinitrine-based medicines
* Recent neurosurgery or traumatic brain injury
* Previous DDAVP or hypertonic fluid administration for the current episode of severe hyponatremia
* SNa increased by 5 mmol or more between admission at hospital and randomisation (H0)
* Known contraindication to DDAVP

  * Allergy
  * Syndrome of inappropriate antidiuretic hormone secretion (SIADH)
  * History of unstable angina and/or known or suspected heart failure.
  * Willebrand disease type IIB
* Severe previous neurologic disability (Glasgow Outcome Scale: GOS < 3)
* Diabetes insipidus receiving DDAVP treatment
* Moribund state (patient likely to die within 24h)
* Need for invasive mechanic ventilation
* Enrolment to another interventional study (clinical trial on medicinal product, medical device and interventional research involving human participants not concerning health product)
* Pregnancy or breastfeeding
* Subject deprived of freedom, subject under a legal protective measure
* No affiliation to any health insurance system
* Refusal to participate to the study (patient or legal representative or family member or close relative if present)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
reduced occurrence of overcorrection of serum sodium concentration (SNa) in the first 48 hours after randomization | 48 hours after the randomization
  proportion of patients with SNa level overcorrection : any risk factor: SNa increase > 6 mmol/L in less than H24, or >12 mmol/L in less than H48. Without risk factor: SNa increase > 10 mmol/L in less than H24, or > 18 mmol/L in less than H48

SECONDARY OUTCOMES:
the reversal of acute neurological symptoms in patients with neurological symptoms at inclusion | 6 hours after the randomization
  proportion of patients with neurological symptoms at inclusion and who subsequently have a normal Glasgow Coma Scale at H6
ICU and hospital length of stay | ICU or hospital discharge
  length of ICU and hospital stay
survival | death after randomization
  time to death after inclusion
the occurrence of central pontine myelinolysis diagnosed on clinical and MRI criteria | 15 days after randomization
  proportion of patients with the occurrence of central pontine myelinolysis diagnosed on clinical and MRI criteria at day 15 (or earlier if clinically justified)
the occurrence of any (pontine or extrapontine) osmotic demyelination as assessed by brain MRI | 15 days after randomization
  proportion of patients with any (pontine or extrapontine), symptomatic or not, osmotic demyelination as assessed by brain MRI at day 15 (or earlier if clinically justified)
on the percentage of patients with neurological symptoms at inclusion and reaching the initial goal of rapid partial pre-defined correction of SNa level | 6 hours after the randomization
  proportion of patients with neurological symptoms with an increase of 5.0 mmol/L or more of SNa from inclusion to H6
the urine output between H0 and H6 | 6 hours after the randomization
  urine output between H0 and H6
the urine output between H6 and H12 | 12 hours after the randomization
  urine output between H6 and H12
the urine output between H12 and H24 | 24 hours after the randomization
  urine output between H12 and H24
the urine output between H24 and H48 | 48 hours after the randomization
  urine output between H24 and H48
the urine osmolality between H0 and H6 | 6 hours after the randomization
  urine osmolality between H0 and H6
the urine osmolality between H6 and H12 | 12 hours after the randomization
  urine osmolality between H6 and H12
the urine osmolality between H12 and H24 | 24 hours after the randomization
  urine osmolality between H12 and H24
the urine osmolality between H24 and H48 | 48 hours after the randomization
  urine osmolality between H24 and H48
SNa level correction rate between H0 and H24 | 24 hours after the randomization
  slope of the SNa increase between H0 and H24
SNa level correction rate between H0 and H48 | 48 hours after the randomization
  slope of the SNa increase between H0 and H48
the maximal change of SNa level between H0 and H24 | 24 hours after the randomization
  maximum change of SNa from baseline between H0 and H24
the maximal change of SNa level between H0 and H48 | 48 hours after the randomization
  maximum change of SNa from baseline between H0 and H48
amount of hypotonic fluids administration | 24 hours after the randomization
  total amount of intravenous hypotonic fluids administered between H0 and H24
amount of hypotonic fluids administration | 48 hours after the randomization
  total amount of intravenous hypotonic fluids administered between H0 and H48
amount of sodium and potassium administered between H0 and H24 | 24 hours after the randomization
  total amount of sodium and potassium administered between H0 and H24
amount of sodium and potassium administered between H0 and H48 | 48 hours after the randomization
  total amount of sodium and potassium administered between H0 and H48
the occurrence of any new neurological sign in relation with hyponatremia in patients with a normal neurological exam at inclusion or on the reappearance of any neurological sign in relation with hyponatremia after inclusion | 28 days after randomization
  proportion of patients with seizures, stupor or sign of brain herniation appearing or reappearing after inclusion
the occurrence of excessive re-lowering of sodium | 48 hours after the randomization
  Occurrence of a reduction of SNa of 5.0 mmol/L or more from inclusion between H0 and H48

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Médecine Intensive et Réanimation - Centre Hospitalier Universitaire Amiens-Picardie, Amiens
  - Médecine Intensive et Réanimation - Hôpital Avicenne, Bobigny
  - Réanimation Polyvalente - Hôpital Jean Verdier, Bondy
  - Médecine Intensive et Réanimation - Hôpital Louis Mourier, Colombes
  - Réanimation Polyvalente et Surveillance continue - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - Médecine Intensive et Réanimation - Hôpital Henri Mondor, Créteil
  - Médecine Intensive et Réanimation - Hôpital François Mitterand, Dijon
  - Réanimation Polyvalente - Centre Hospitalier Départemental Vendée, La Roche-sur-Yon
  - Réanimation Médicale - Hôpital de Longjumeau, Longjumeau
  - Médecine Intensive et Réanimation - Hôpital de la Pitié Salpêtrière, Paris
  - Médecine Intensive Réanimation - Hôpital Delafontaine, Saint-Denis
  - Réanimation Polyvalente - Hôpital Foch, Suresnes

IPD SHARING:
Plan to Share IPD: No